CLINICAL TRIAL: NCT03046732
Title: Reducing Barriers in Access to Kidney Transplantation: Implementing the "Explore Transplant" Education Program to Increase Patient Knowledge and to Facilitate Informed Decision Making- A Pilot Study
Brief Title: Implementing "Explore Transplant"- A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Istvan Mucsi, Transplant Nephrologist, University Health Network, Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-5314-AE
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Endstage Kidney Disease
Keywords: Kidney Transplant Education; Transplant Readiness; Living Donor Kidney Transplant; Chronic Kidney Disease; End Stage Kidney Disease; Renal Replacement Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Explore Transplant Ontario (Experimental): Intervention 'Implementing "Explore Transplant" Education'
  Interventions: Other: Implementing "Explore Transplant" Education
- Control (No Intervention): The control arm (Usual Treatment) is at the Toronto General Hospital dialysis center.

INTERVENTIONS:
Other: Implementing "Explore Transplant" Education — The "Explore Transplant Ontario" (ETO) education program
  Arms: Explore Transplant Ontario

SUMMARY:
Patients with End Stage Kidney Disease (ESKD) require Renal Replacement Therapy (RRT) in order to survive, be it dialysis or kidney transplantation (KT). Of the two modalities, KT has been associated with better quality of life (QOL) [1-3], reduced morbidity and mortality[4, 5], and reduced healthcare costs[6]. Studies in the US have shown that patients receiving tailored transplant education were more likely to complete the transplant evaluation [9, 14, 15]. For instance, patients receiving the Explore Transplant (ET) education program designed by Dr. Waterman, were more knowledgeable about KT and more likely to complete KT evaluation than control patients. Currently, there is a lack of standardized KT education in Ontario. Traditional approaches have been insufficient in providing the necessary education and information to enable patients to make an informed decision about their care. To address this issue, the study will assess the impact of kidney transplant related education using the Explore Transplant Ontario (ETO) education program on kidney transplant-related knowledge and on readiness to consider KT, readiness to consider living donor KT, and wait list/referral rates in patients undergoing maintenance hemodialysis.

In order to comprehensively measure this impact, 5 variables will be explored.

1. Readiness to consider DDKT
2. Readiness to consider LDKT
3. KT related knowledge in patients
4. Proportion of patients waitlisted or undergoing KT workup at 6 and 12 months after administration of ETO
5. Proportion of patients who have identified at least one potential living donor at 6 and 12 months after administration of ETO

The hypotheses are as follows:

1. Readiness to consider DDKT will be higher in the "intervention" group compared to the "control" group at follow up.
2. Readiness to consider LDKT will be higher in the "intervention" group compared to the "control" group at follow up.
3. The KT related knowledge of the patients will be higher in the "intervention" group compared to the "control" group at follow up.
4. The proportion of patients waitlisted or undergoing KT workup at 6 and 12 month after the KT education will be higher in the "intervention" group compared to the "control" group.
5. The proportion of patients who have at least one potential living donor at 6 and 12 month after the KT education will be higher in the "intervention" group compared to the "control" group.

DETAILED DESCRIPTION:
ESKD impairs quality of life (QOL)QoL and leads to increased morbidity and premature mortality. In addition, healthcare costs for ESKD amounted to $1.3 billion in Canada in 2000 [22]. KT has clear survival [4] and QOL [1-3], and economic benefits [6]. Studies in the US documented that tailored education improves KT knowledge and enhances access to KT and LDKT [14, 23-26]. Current education materials and teaching for KT candidates in Ontario are not based on theoretical foundations or on research evidence. This has resulted in gaps in transplant education in Ontario and has been unable to meet the needs of the patients. By building upon research data from the US we aim to implement a culturally sensitive patient education tool that will address the current needs as well as reduce barriers whereby enhancing access to KT.

This project will increase KT knowledge among health care professionals and among patients. We will establish ongoing support for the participating nephrology centers. This will also increase KT knowledge in patients and families and enhance access to KT. The ultimate goal is to improve health outcomes and QOL by reducing barriers to KT and LDKT and to help patients and families make informed treatment decisions.

The Explore Transplant Ontario (ETO) is a parallel, non-randomized, controlled pilot study exploring the impact of an educational intervention designed to increase knowledge about kidney transplantation (KT) and readiness to consider KT. For this pilot study we will utilize a convenience sample of stable patients on hemodialysis in two large dialysis units. The "intervention" will be administered at the hemodialysis unit at Humber River Hospital; the "control" group will be recruited from the hemodialysis unit at Toronto General Hospital. Currently around 500 patients are being treated with maintenance hemodialysis in both dialysis units, with an estimate that about 300 of these patients will fulfill our inclusion criteria.

The estimated study period will be 21 months. Baseline study recruitment will occur over a period of 3 months at each of the participating dialysis centers. Data management, follow-up, and analysis will take place over the subsequent 18 months.The study recruitment period has about 60 business days and as such, recruitment rate is estimated at 5-6 patients per day of screening.

The entire study will take place over 4 distinct stages

Stage 1:

Baseline data collection will be conducted at both dialysis centers

Stage 2:

A full day training will be organized to train a selected group of dialysis nurses. This group will act as a group of clinical experts and help facilitate training and use of the ETO amongst the other health care practitioners.

Stage 3:

Following the training session, ETO will be implemented at the hemodialysis unit at Humber River Hospital as the "intervention" arm and at the Toronto General Hospital as the "control" arm. It is estimated that 300 of the hemodialysis patients will fulfill the inclusion criteria, resulting in an enrollment of 150 patients in each study arm.

Stage 4:

The study duration will take approximately 21 months to accomplish. Baseline recruitment will occur over a period of 3 months at each participating dialysis centers, estimating 5-6 patients per day of screening. Data management, follow-up, and analysis will take place over the subsequent 18 months.

Statistical Analysis Plan:

Categorical variables ("early versus "late" stage of readiness, high versus low knowledge) will be compared using logistic regression models (knowledge or readiness stage as the dependent variable; exposure to ETO education is the primary explanatory variable). Continuous knowledge score will also be analyzed in linear regression models (score as the dependent variable, exposure to ET as the primary explanatory variable). These analyses will then be adjusted for age, gender, education, ethnicity/race and comorbidity.

Chi-square test will be used to compare the proportions of patients on KT waiting list and under KT evaluation in the control versus the intervention group, both at baseline and at the 3 month follow up.

Baseline data about the proportion of patients on the KT waiting list and under KT evaluation in participating dialysis centers will be collected at the participating dialysis units.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, < 80 years
* Patients undergoing maintenance hemodialysis for more than 3 months
* Able to understand English at a grade 5 level
* Those willing and able to provide informed consent

Exclusion Criteria:

* Patients with severe acute illness or condition that hampers questionnaire completion
* Dementia indicated in the medical record, indicated by the managing healthcare team
* Dialysis initiation between 0-90 days prior to enrollment
* Current, active malignancy or a history of malignancy within 2 years of successful treatment
* Current active chronic infection that is an absolute contraindication to kidney transplantation
* Unwilling or unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in "early stages" of kidney transplant readiness | An average of 1 year and a half

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Mucsi, Principal Investigator — Toronto General Hospital
Locations (2):
- Canada (2):
  - Humber River Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kovacs AZ, Molnar MZ, Szeifert L, Ambrus C, Molnar-Varga M, Szentkiralyi A, Mucsi I, Novak M. Sleep disorders, depressive symptoms and health-related quality of life--a cross-sectional comparison between kidney transplant recipients and waitlisted patients on maintenance dialysis. Nephrol Dial Transplant. 2011 Mar;26(3):1058-65. doi: 10.1093/ndt/gfq476. Epub 2010 Aug 4. PMID 20685829
- [Background] Kostro JZ, Hellmann A, Kobiela J, Skora I, Lichodziejewska-Niemierko M, Debska-Slizien A, Sledzinski Z. Quality of Life After Kidney Transplantation: A Prospective Study. Transplant Proc. 2016 Jan-Feb;48(1):50-4. doi: 10.1016/j.transproceed.2015.10.058. PMID 26915842
- [Background] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Background] Tennankore KK, Kim SJ, Baer HJ, Chan CT. Survival and hospitalization for intensive home hemodialysis compared with kidney transplantation. J Am Soc Nephrol. 2014 Sep;25(9):2113-20. doi: 10.1681/ASN.2013111180. Epub 2014 May 22. PMID 24854268
- [Background] Eggers P. Comparison of treatment costs between dialysis and transplantation. Semin Nephrol. 1992 May;12(3):284-9. No abstract available. PMID 1615249
- [Background] Patzer RE, Plantinga L, Krisher J, Pastan SO. Dialysis facility and network factors associated with low kidney transplantation rates among United States dialysis facilities. Am J Transplant. 2014 Jul;14(7):1562-72. doi: 10.1111/ajt.12749. Epub 2014 May 29. PMID 24891272
- [Background] Schold JD, Srinivas TR, Kayler LK, Meier-Kriesche HU. The overlapping risk profile between dialysis patients listed and not listed for renal transplantation. Am J Transplant. 2008 Jan;8(1):58-68. doi: 10.1111/j.1600-6143.2007.02020.x. Epub 2007 Nov 2. PMID 17979999
- [Background] Waterman AD, Peipert JD, Hyland SS, McCabe MS, Schenk EA, Liu J. Modifiable patient characteristics and racial disparities in evaluation completion and living donor transplant. Clin J Am Soc Nephrol. 2013 Jun;8(6):995-1002. doi: 10.2215/CJN.08880812. Epub 2013 Mar 21. PMID 23520044
- [Background] Vamos EP, Csepanyi G, Zambo M, Molnar MZ, Rethelyi J, Kovacs A, Marton A, Nemeth Z, Novak M, Mucsi I. Sociodemographic factors and patient perceptions are associated with attitudes to kidney transplantation among haemodialysis patients. Nephrol Dial Transplant. 2009 Feb;24(2):653-60. doi: 10.1093/ndt/gfn660. Epub 2008 Nov 30. PMID 19047018
- [Background] Salter ML, Orandi B, McAdams-DeMarco MA, Law A, Meoni LA, Jaar BG, Sozio SM, Kao WH, Parekh RS, Segev DL. Patient- and provider-reported information about transplantation and subsequent waitlisting. J Am Soc Nephrol. 2014 Dec;25(12):2871-7. doi: 10.1681/ASN.2013121298. Epub 2014 Aug 28. PMID 25168028
- [Background] Olbrisch ME, Benedict SM, Haller DL, Levenson JL. Psychosocial assessment of living organ donors: clinical and ethical considerations. Prog Transplant. 2001 Mar;11(1):40-9. doi: 10.1177/152692480101100107. PMID 11357556
- [Background] Kasiske BL. The evaluation of prospective renal transplant recipients and living donors. Surg Clin North Am. 1998 Feb;78(1):27-39. doi: 10.1016/s0039-6109(05)70632-0. PMID 9531933
- [Background] Rodrigue JR, Paek MJ, Egbuna O, Waterman AD, Schold JD, Pavlakis M, Mandelbrot DA. Making house calls increases living donor inquiries and evaluations for blacks on the kidney transplant waiting list. Transplantation. 2014 Nov 15;98(9):979-86. doi: 10.1097/TP.0000000000000165. PMID 24825528
- [Background] Rodrigue JR, Pavlakis M, Egbuna O, Paek M, Waterman AD, Mandelbrot DA. The "House Calls" trial: a randomized controlled trial to reduce racial disparities in live donor kidney transplantation: rationale and design. Contemp Clin Trials. 2012 Jul;33(4):811-8. doi: 10.1016/j.cct.2012.03.015. Epub 2012 Apr 3. PMID 22510472
- [Background] Weng FL, Brown DR, Peipert JD, Holland B, Waterman AD. Protocol of a cluster randomized trial of an educational intervention to increase knowledge of living donor kidney transplant among potential transplant candidates. BMC Nephrol. 2013 Nov 19;14:256. doi: 10.1186/1471-2369-14-256. PMID 24245948
- [Background] Waterman AD, Robbins ML, Paiva AL, Hyland SS. Kidney patients' intention to receive a deceased donor transplant: development of stage of change, decisional balance and self-efficacy measures. J Health Psychol. 2010 Apr;15(3):436-45. doi: 10.1177/1359105309351248. PMID 20348364
- [Background] Terasaki PI, Cecka JM, Gjertson DW, Takemoto S. High survival rates of kidney transplants from spousal and living unrelated donors. N Engl J Med. 1995 Aug 10;333(6):333-6. doi: 10.1056/NEJM199508103330601. PMID 7609748
- [Background] Waterman AD, Stanley SL, Covelli T, Hazel E, Hong BA, Brennan DC. Living donation decision making: recipients' concerns and educational needs. Prog Transplant. 2006 Mar;16(1):17-23. doi: 10.1177/152692480601600105. PMID 16676669
- [Background] Pradel FG, Mullins CD, Bartlett ST. Exploring donors' and recipients' attitudes about living donor kidney transplantation. Prog Transplant. 2003 Sep;13(3):203-10. doi: 10.1177/152692480301300307. PMID 14558635
- [Background] Zelmer JL. The economic burden of end-stage renal disease in Canada. Kidney Int. 2007 Nov;72(9):1122-9. doi: 10.1038/sj.ki.5002459. Epub 2007 Aug 15. PMID 17700643
- [Background] Waterman AD, Rodrigue JR, Purnell TS, Ladin K, Boulware LE. Addressing racial and ethnic disparities in live donor kidney transplantation: priorities for research and intervention. Semin Nephrol. 2010 Jan;30(1):90-8. doi: 10.1016/j.semnephrol.2009.10.010. PMID 20116653
- [Background] Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, McGuire R, Bonhage B, Senga M, Ephraim P, Evans KE, Falcone B, Troll MU, Depasquale N, Powe NR. Protocol of a randomized controlled trial of culturally sensitive interventions to improve African Americans' and non-African Americans' early, shared, and informed consideration of live kidney transplantation: the Talking About Live Kidney Donation (TALK) Study. BMC Nephrol. 2011 Jul 8;12:34. doi: 10.1186/1471-2369-12-34. PMID 21736762
- [Background] DePasquale N, Ephraim PL, Ameling J, Lewis-Boyer L, Crews DC, Greer RC, Rabb H, Powe NR, Jaar BG, Gimenez L, Auguste P, Jenckes M, Boulware LE. Selecting renal replacement therapies: what do African American and non-African American patients and their families think others should know? A mixed methods study. BMC Nephrol. 2013 Jan 14;14:9. doi: 10.1186/1471-2369-14-9. PMID 23317336
- [Background] Ephraim PL, Powe NR, Rabb H, Ameling J, Auguste P, Lewis-Boyer L, Greer RC, Crews DC, Purnell TS, Jaar BG, DePasquale N, Boulware LE. The providing resources to enhance African American patients' readiness to make decisions about kidney disease (PREPARED) study: protocol of a randomized controlled trial. BMC Nephrol. 2012 Oct 12;13:135. doi: 10.1186/1471-2369-13-135. PMID 23057616
- [Background] Hall KL, Robbins ML, Paiva A, Knott JE, Harris L, Mattice B. Donation intentions among African American college students: decisional balance and self-efficacy measures. J Behav Med. 2007 Dec;30(6):483-95. doi: 10.1007/s10865-007-9121-8. Epub 2007 Aug 3. PMID 17674183
- [Background] Waterman AD, Dew MA, Davis CL, McCabe M, Wainright JL, Forland CL, Bolton L, Cooper M. Living-donor follow-up attitudes and practices in U.S. kidney and liver donor programs. Transplantation. 2013 Mar 27;95(6):883-8. doi: 10.1097/TP.0b013e31828279fd. PMID 23388736
- [Background] Waterman AD, Robbins ML, Paiva AL, Peipert JD, Davis LA, Hyland SS, Schenk EA, Baldwin KA, Amoyal NR. Measuring kidney patients' motivation to pursue living donor kidney transplant: development of stage of change, decisional balance and self-efficacy measures. J Health Psychol. 2015 Feb;20(2):210-21. doi: 10.1177/1359105313501707. Epub 2013 Oct 22. PMID 24155194
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Christensen, A.J., et al., Quality of life in end-stage renal disease: Influence of renal transplantation. Clin Transplant, 1989. 3: p. 46-53
- [Background] Information, C.I.H.I., 2014 CORR Report: Treatment of End-Stage Organ Failure in Canada, 2003 to 2012. 2014.
- [Background] Report, T.-H.T., We ask because we care- The Tri-Hospital + TPH Health Equity Data Collection Research Project Report. 2013: p. 51.
- See also: Canada, S. Classificiation of population group 2009 [cited 2015 August 5th, 2015] — https://www.statcan.gc.ca/en/concepts/definitions/previous/preethnicity